CLINICAL TRIAL: NCT04502524
Title: A Scalable e-Health Smoking Cessation Intervention for Socioeconomically Disadvantaged Veterans
Brief Title: Website Smoking Cessation Intervention for the Promotion of Smoking Cessation in Low-Income Veterans
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Jaimee Heffner, Associate Professor, Fred Hutchinson Cancer Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: RG1007109; NCI-2020-05587 (Registry Identifier: NCI / CTRP); R21CA236980 (NIH); 10097 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2020-07-30; First posted 2020-08-06 (Actual); Results first posted 2023-04-07 (Actual); Last update posted 2023-04-07 (Actual); Status verified 2023-03

CONDITIONS: Cigarette Smoking-Related Carcinoma
MeSH Terms: interventions — Smoking Devices; Standard of Care; Practice Guidelines as Topic; Health Promotion; Educational Status

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm I (New website program, handout, text message) (Experimental): Participants complete the new website smoking cessation program which provides values driven, mindfulness based coping skills and utilizes non-judgmental acceptance of uncomfortable internal states like cravings. Participants will also receive text messages consisting of motivational messages and reminders to use the program. At the end of the program, participants receive an email with all session handouts and available resources provided by the VA for continued support for smoking cessation.
  Interventions: Behavioral: Smoking Cessation Intervention (New website); Behavioral: Health Education; Other: Health Promotion and Education; Other: Questionnaire Administration
- Arm II (Standard care VA website, handout, text message) (Active Comparator): Participants use the standard of care website, which provides educational materials about cessation treatments, tools to cope with urges and relapse, how to stay motivated, and brief tips on coping with physical and mental health problems. Participants also receive text messages consisting of motivational messages and reminders to use the program. At the end of the program, participants receive an email with a handout of available resources provided by the VA for continued support for smoking cessation.
  Interventions: Behavioral: Smoking Cessation Intervention (Standard of care website); Behavioral: Health Education; Other: Health Promotion and Education; Other: Questionnaire Administration

INTERVENTIONS:
Behavioral: Smoking Cessation Intervention (New website) — Complete the new website smoking cessation program
  Other Names: Smoking and Tobacco Use Cessation Interventions
  Arms: Arm I (New website program, handout, text message)
Behavioral: Smoking Cessation Intervention (Standard of care website) — Complete the standard of care website smoking cessation intervention
  Other Names: standard of care; standard therapy; best practice
  Arms: Arm II (Standard care VA website, handout, text message)
Behavioral: Health Education — Receive information about the cost of smoking, benefits of quitting, ways to prepare for quitting, ways to handle triggers and withdrawal symptoms, and available medications to help with quitting. And will receive additional resources available at the VA handout via email at the end of the study.
Other: Health Promotion and Education — Receive motivational and reminder text messages
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This phase I trial studies how well a new electronic (e)-health smoking cessation program (called Vet Flexiquit) works in promoting smoking cessation in low-income veterans who may or may not be ready to quit smoking. The study will compare the new website smoking cessation program to the current standard care website smoking cessation program offered by the Veterans Administration (VA). Both website interventions will be accompanied by a text messaging program that includes: (1) motivational messages, and (2) reminders to use the assigned program. Both of the website interventions can help smokers quit or cut back on how much they smoke, thus dramatically reducing their chances of developing tobacco-related health conditions.

DETAILED DESCRIPTION:
OUTLINE: Participants are randomized to 1 of 2 arms.

ARM I: Participants use the new website smoking cessation program, which provides values driven, mindfulness based coping skills and utilizes non-judgmental acceptance of uncomfortable internal states like cravings. Participants also receive text messages consisting of motivational messages and reminders to use the program. At the end of the program, participants receive an email with handouts and available resources provided by the VA for continued support for smoking cessation.

ARM II: Participants use the VA standard of care website, which provides educational materials about cessation treatments, tools to cope with urges and relapse, how to stay motivated, and brief tips on coping with physical and mental health problems. Participants also receive text messages consisting of motivational messages and reminders to use the program. At the end of the program, participants receive an email with a handout of available resources provided by the VA for continued support for smoking cessation.

After study randomization, participants are followed up at 1 and 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be a US veteran
* Participants must be low-income, as defined by falling below Veterans Health Administration (VHA) national income threshold for no-cost healthcare
* Participants must be a current smoker, averaging at least 5 cigarettes/day for the last 30 days
* Participants must have weekly internet access for the next 3 months
* Participants must self-report current use of a personal email address to receive the link to their assigned web site
* Participants must self-report being willing to complete all study activities
* Participants must be willing to receive study-related text messages

Exclusion Criteria:

* Currently taking part in any other smoking cessation treatment such as the nicotine patch, nicotine gum, Zyban, in-person counseling, telephone counseling, using a web-based or app-based cessation program
* Have recent (past 30 days) substance use disorder, suicidal ideation, or psychiatric hospitalization
* Previous participation in the treatment development stage of the new smoking cessation website program
* Prior use of the SmokefreeVET web site
* Member of the same household as another research participant
* Woman who is pregnant or breastfeeding, or planning to become pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2021-02-03 (Actual); Primary Completion 2022-01-28 (Actual); Study Completion 2022-01-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jaimee Heffner, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Bedford VA Research Corporation, Inc., Bedford, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Heffner JL, Kelly MM, Reilly ED, Reece SG, Claudio T, Serfozo E, Baker K, Watson NL, Karekla M. An Avatar-Led Web-Based and SMS Text Message Smoking Cessation Program for Socioeconomically Disadvantaged Veterans: Pilot Randomized Controlled Trial. JMIR Form Res. 2023 Apr 14;7:e44503. doi: 10.2196/44503. PMID 37058346

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Fifty-three participants were eligible and enrolled in the study. The final sample comprised 49 participants who were randomized between February 3, 2021 and October 22, 2021.
Pre-assignment Details: Four participants who were enrolled in the study were not randomized because they were lost to follow-up (n=3) or they withdrew (n=1) prior to randomization.
Period: Overall Study
Arm/Group | Arm I (New Website Program, Handout, Text Message) | Arm II (Standard Care VA Website, Handout, Text Message)
Started | 25 | 24
Completed | 18 | 20
Not Completed | 7 | 4

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (New Website Program, Handout, Text Message) | Arm II (Standard Care VA Website, Handout, Text Message) | Total
Number analyzed (Participants) | 25 | 24 | 49
Age, Continuous [Mean (Full Range); unit: years] | 47.9 [26 to 74] | 54.8 [27 to 84] | 51.3 [26 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 7 | 12
  Male | 20 | 17 | 37
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 2
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 2 | 4
  White | 19 | 20 | 39
  More than one race | 2 | 2 | 4
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 25 | 24 | 49
Fagerström Test for Nicotine Dependence (FTND) [Mean (Full Range); unit: units on a scale] — The 6-item Fagerström Test for Nicotine Dependence (FTND) was used to assess degree of physical dependence on nicotine. Scale range is from 0-10. Higher scores indicate higher dependence.
  units on a scale | 4.3 [0.0 to 8] | 4.2 [0.0 to 7] | 4.3 [0.0 to 8]
Contemplation Ladder [Mean (Standard Deviation); unit: units on a scale] — Range is from 0-10. Higher scores indicate greater readiness to quit.
  units on a scale | 8.0 (2.3) | 7.8 (2.1) | 7.9 (2.2)

OUTCOME MEASURES:

1. Primary Outcome: Satisfaction With Assigned Treatment
Description: Satisfaction ratings regarding the usefulness of specific components of the website program, user comments and suggestions for improvement, presented descriptively. Treatment satisfaction items are reported on a Likert-type scale, with response choices ranging from "not at all satisfied" to "very satisfied". Will dichotomize values at a threshold of "somewhat satisfied" or higher. We tested for differences between arms using a Fisher's Exact test.
Time Frame: At 3 months post-randomization
Population: All survey respondents
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (New Website Program, Handout, Text Message) | Arm II (Standard Care VA Website, Handout, Text Message)
Number analyzed (Participants) | 17 | 19
Participants
  Not At All/A Little | 0 | 1
  Somewhat/Mostly/Very Much | 17 | 18
Statistical Analysis 1: Comparison: Arm I (New Website Program, Handout, Text Message) vs Arm II (Standard Care VA Website, Handout, Text Message); For overall satisfaction, a reliable estimate could not be calculated using a logistic regression model as all the responses were the same in the Vet Flexiquit arm. We calculated the p-value using the Fisher's exact test; Test type: Other; p = .999, Fisher Exact

2. Primary Outcome: Number of Server-recorded Logins to Assigned Website
Description: Will use negative binomial regression with adjustment for the stratification variable and baseline readiness to quit (high versus low) to compare treatment effects on the count outcome number of logins. There were no potential confounders to adjust for.
Time Frame: At 3 months
Population: All survey respondents.
Measure: Mean (Standard Deviation); unit: Count of number of times logged in
Arm/Group | Arm I (New Website Program, Handout, Text Message) | Arm II (Standard Care VA Website, Handout, Text Message)
Number analyzed (Participants) | 17 | 19
Count of number of times logged in | 3.7 (3.6) | 3.2 (4.1)
Statistical Analysis 1: Comparison: Arm I (New Website Program, Handout, Text Message) vs Arm II (Standard Care VA Website, Handout, Text Message); Test type: Other; p = 0.852, Regression, negative binomial; Slope = 0.05, 95% CI 2-sided [-0.46 to 0.56]

3. Primary Outcome: Duration of Website Use (Days Since First Login)
Description: Will use negative binomial regression with adjustment for the stratification variable baseline readiness to quit (high versus low) to compare treatment groups on the secondary acceptability outcome of duration of site usage (number of days elapsed from first to last use). There were no confounders to adjust for.
Time Frame: At 3 months
Population: All randomized participants.
Measure: Mean (Standard Deviation); unit: Days since first login
Arm/Group | Arm I (New Website Program, Handout, Text Message) | Arm II (Standard Care VA Website, Handout, Text Message)
Number analyzed (Participants) | 17 | 19
Days since first login | 18.7 (27.3) | 26.7 (47.2)
Statistical Analysis 1: Comparison: Arm I (New Website Program, Handout, Text Message) vs Arm II (Standard Care VA Website, Handout, Text Message); Test type: Other; p = 0.451, Regression, negative binomial; Slope = -0.44, 95% CI 2-sided [-1.60 to 0.71]

4. Secondary Outcome: Number of Quit Attempts
Description: Will use a negative binomial model with adjustment for the stratification variable and baseline readiness to quit (high versus low) to compare the count outcome number of quit attempts between arms. There were no confounders to address for.
Time Frame: At 3 months
Population: All survey respondents.
Measure: Mean (Standard Deviation); unit: Number of quit attempts
Arm/Group | Arm I (New Website Program, Handout, Text Message) | Arm II (Standard Care VA Website, Handout, Text Message)
Number analyzed (Participants) | 18 | 19
Number of quit attempts | 1.7 (1.1) | 3.2 (6.7)
Statistical Analysis 1: Comparison: Arm I (New Website Program, Handout, Text Message) vs Arm II (Standard Care VA Website, Handout, Text Message); Test type: Other; p = 0.508, Regression, negative binomial; Slope = -0.73, 95% CI 2-sided [-1.46 to 0.003]

5. Secondary Outcome: Cotinine-confirmed, Self-reported Abstinence From Smoking
Description: Will use a logistic regression model with adjustment for the stratification variable and baseline readiness to quit (high versus low) to compare smoking abstinence between arms. There were no confounders to adjust for. Missing responses were considered as continued smokers.
Time Frame: In the 7 days prior to the 3-month follow up
Population: All survey respondents.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (New Website Program, Handout, Text Message) | Arm II (Standard Care VA Website, Handout, Text Message)
Number analyzed (Participants) | 25 | 24
Participants | 3 | 4
Statistical Analysis 1: Comparison: Arm I (New Website Program, Handout, Text Message) vs Arm II (Standard Care VA Website, Handout, Text Message); Test type: Other; p = 0.602, Regression, Logistic; Odds Ratio (OR) = 0.65, 95% CI 2-sided [0.13 to 3.32]

6. Secondary Outcome: Cotinine-confirmed, Self-reported Abstinence From Smoking
Description: Will use a logistic regression model with adjustment for the stratification variable and baseline readiness to quit (high versus low) to compare smoking abstinence between arms. There were no confounders to adjust for. Missing responses were considered continued smokers.
Time Frame: In the 30 days prior to the 3-month follow up
Population: All survey respondents.
Measure: Number; unit: participants
Arm/Group | Arm I (New Website Program, Handout, Text Message) | Arm II (Standard Care VA Website, Handout, Text Message)
Number analyzed (Participants) | 25 | 24
participants | 3 | 3
Statistical Analysis 1: Comparison: Arm I (New Website Program, Handout, Text Message) vs Arm II (Standard Care VA Website, Handout, Text Message); Test type: Other; p = 0.941, Regression, Logistic; Odds Ratio (OR) = 0.94, 95% CI 2-sided [0.17 to 5.29]

7. Secondary Outcome: Self-reported Abstinence From All Nicotine and Tobacco Products (Except Nicotine Replacement Therapy)
Description: Will use a logistic regression model with adjustment for the stratification variable and baseline readiness to quit (high versus low) to compare smoking abstinence between arms. There were no confounders to adjust for. The missing responses were considered continued smokers.
Time Frame: In the 7 days prior to the 3-month follow up
Measure: Number; unit: participants
Arm/Group | Arm I (New Website Program, Handout, Text Message) | Arm II (Standard Care VA Website, Handout, Text Message)
Number analyzed (Participants) | 24 | 24
participants | 2 | 3
Statistical Analysis 1: Comparison: Arm I (New Website Program, Handout, Text Message) vs Arm II (Standard Care VA Website, Handout, Text Message); Test type: Other; p = 0.612, Regression, Logistic; Odds Ratio (OR) = 0.61, 95% CI 2-sided [0.09 to 4.12]

8. Secondary Outcome: Change in Readiness to Quit
Description: Will be assessed by the Contemplation Ladder on a scale from 0 (no thought about quitting) to 10 (taking action to quit). Will calculate change score as follow-up minus baseline score and use a linear regression model with adjustment for the baseline value of the measure of interest and for the stratification variable and baseline readiness to quit (high versus low) to compare between study arms. There were no confounders to adjust for.
Time Frame: Baseline up to 3-month follow-up
Population: All survey respondents.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm I (New Website Program, Handout, Text Message) | Arm II (Standard Care VA Website, Handout, Text Message)
Number analyzed (Participants) | 18 | 19
score on a scale | -0.4 (3.3) | -0.5 (3.6)
Statistical Analysis 1: Comparison: Arm I (New Website Program, Handout, Text Message) vs Arm II (Standard Care VA Website, Handout, Text Message); Test type: Other; p = 0.504, Regression, Linear; Slope = 0.56, 95% CI 2-sided [-1.13 to 2.26]

9. Secondary Outcome: Change in Acceptance of Smoking Triggers
Description: Will be assessed by the Avoidance and Inflexibility Scale (AIS) on a scale ranging from 0 (never/not at all) to 4 (always/very much/extensively). Will calculate change score as follow-up minus baseline score and use a linear regression model with adjustment for the baseline value of the measure of interest and for the stratification variable and baseline readiness to quit (high versus low) to compare between study arms. There were no confounders to adjust for. This is the AIS Feelings score change.
Time Frame: Baseline up to 3-month follow-up
Population: All survey respondents.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm I (New Website Program, Handout, Text Message) | Arm II (Standard Care VA Website, Handout, Text Message)
Number analyzed (Participants) | 18 | 20
score on a scale | 0.4 (0.6) | 0.3 (0.8)
Statistical Analysis 1: Comparison: Arm I (New Website Program, Handout, Text Message) vs Arm II (Standard Care VA Website, Handout, Text Message); Test type: Other; p = 0.670, Regression, Linear; Slope = 0.11, 95% CI 2-sided [-0.40 to 0.61]

ADVERSE EVENTS:
Time Frame: 3-months
Description: Volunteered adverse events collected throughout the 3-month follow-up.
Arm/Group | Arm I (New Website Program, Handout, Text Message) | Arm II (Standard Care VA Website, Handout, Text Message)
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/24
Other Adverse Events (participants affected / at risk) | 0/25 | 0/24

LIMITATIONS AND CAVEATS:
The goal was to establish feasibility rather than to detect statistically significant differences between arms. The sample size was small, and follow-ups were limited to short-term outcomes. Some ACT interventions have demonstrated greater effects when evaluated at long-term follow-up. This study was conducted during the COVID-19 pandemic, which represents a unique context. The study design was also impacted by the pandemic, transforming a primarily in-person design to a fully remote one.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-04-15): https://cdn.clinicaltrials.gov/large-docs/24/NCT04502524/Prot_SAP_001.pdf
  • Informed Consent Form (2020-12-18): https://cdn.clinicaltrials.gov/large-docs/24/NCT04502524/ICF_000.pdf